CLINICAL TRIAL: NCT03009370
Title: The Effect of the Ovarian Reserve on the Recurrent Pregnancy Loss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gonca Yetkin Yildirim, MD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KanuniSSSTRH
Record Dates: First submitted 2016-12-18; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Ovarian Reserve; Miscarriage, Recurrent
Keywords: Ovarian reserve, pregnancy loss
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Recurrent miscarriage: RM is defined as three or more pregnancy losses at< 20 weeks of gestation.

SUMMARY:
The purpose of this study is to determine whether ovarian reserve is related to recurrent pregnancy loss

DETAILED DESCRIPTION:
This study will be conducted at the gynecology and infertility department of Kanuni Sultan Süleyman Training and Research Hospital from 2016 to 2017. The approval of the local Institutional Review Board (KAEK/2016.22.31) was obtained in June 2016 and informed consents of all subjects have been prepared. RM is defined as three or more pregnancy losses at <20 weeks of gestation or fetal weight <500 g. Women with history of RM for whom routine workup for RM (chromosomal analyses of both partners; levels of prolactin and TSH; anticardiolipin antibody, lupus anticoagulant, antinuclear antibody, and coagulation studies; and pelvic ultrasonography) is negative are assigned to the RM group. The control group consists of healthy women with no history of RM who are seeking contraception in the center's family planning unit. To keep the power of the study at 80% with an alpha-level of 0.05, a sample size of minumum 60 patients in each group was required.

Demographic data (age,gravidity,parity,pregnancy loss,bmı) ovarian reserve parameters(AMH,FSH,LH,E2,AFC) will be recorded and then two groups will be compared.

Data will be analyzed with the use of medcalc version 16.4.8 by Gökhan Yıldırım. Mean,median,SD,lowest and highest frequency ,and ratio values are used at statistical complementary of data .Quantitative data will be analyzed with the use of the Student t test and the Mann-Whitney U test. A chisquare test will be used for analyses of qualitative data

ELIGIBILITY:
Inclusion Criteria:

* Women with RM between 20-40 years old

Exclusion Criteria:

* Anovulation or PCOS
* Presence of endometrosis by laparoscopy or ultrasonography
* History of ovarian surgery
* Tobacco use
* Systemic chemotherapy
* Pelvic irradition
* Genetic abnormalities
* Irregular menstruel cycle
* family history of premature ovarian failure

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recurrent miscarriage is defined as three or more pregnancy loss at<20 weeks of gestation.The women between 20 -40 years old with history of RM are recruited.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The effect of the ovarian reserve on the recurrent pregnancy loss | up to 6 months
  Venous blood samples will be taken from the antecubital regions of all patients between 8:00 a.m and 9:00 a.m during the early follicular phase (days 2-4) of the menstrual cycle .Serum samples will be stored at -80C and assayed for FSH,LH,E2 and AMH .FSH levels are analyzed by means of an electrochemiluminescence method .The normal range for FSH is 2.5-10 U/L at the early follicular phase. Serum AMH levels will be measured with the use of a human ELİSA kit . The normal range for this assay is 0.05-1.5 ng/ml.In the same morning that the blood tests are performed , the total number of antral follicles measuring 2-10 mm in diameter are evaluated by the operator.A 7.5 -MHz transvaginal probe is used in all examinations.Data will be analyzed with the use of medcalc.

SECONDARY OUTCOMES:
Ovarian reserve tests can be used for the diagnosis of the cause of recurrent pregnancy loss | up to 6 months
  FSH,LH,E2,AMH assesment of at least 86 patients will be analyzed with the use of medcalc . Unıts of measure of FSH,LH,E2 levels are assesed by U/L. The normal range of AMH level is 0.05-1.5ng/ml. Mean ,median ,SD, lowest and highest frequency ,and ratio values are used at statistical complemantary data.Quantitative data are analyzed with the use of the student -t test and Mann-Whitney U test

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Yetkin Yıdırım, MD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Atasever M, Soyman Z, Demirel E, Gencdal S, Kelekci S. Diminished ovarian reserve: is it a neglected cause in the assessment of recurrent miscarriage? A cohort study. Fertil Steril. 2016 May;105(5):1236-1240. doi: 10.1016/j.fertnstert.2016.01.001. Epub 2016 Jan 21. PMID 26806685
- Available data/document: Study Protocol — http://www.ncbi.nlm.nih.gov/pubmed/26806685